CLINICAL TRIAL: NCT06259435
Title: Modulating Energy Density in Time-Restricted Eating
Acronym: MEDITRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Candida Rebello, Assistant Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PBRC-2023-049
Record Dates: First submitted 2024-01-26; First posted 2024-02-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Insulin Resistance; Body Weight
MeSH Terms: conditions — Insulin Resistance; Body Weight

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to receive a diet low in energy density or the usual diet.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects will be randomly assigned to one of two groups. Except for the Director of the Metabolic Kitchen and the dietitians assigned to the study, all other researchers conducting the study will be blinded to the treatment group assignment of subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low energy dense diet (Experimental): Subjects will be required to follow time-restricted eating and receive a diet low in energy density
  Interventions: Behavioral: Low-energy dense diet
- Usual diet (Active Comparator): Subjects will be required to follow time-restricted eating and receive the usual diet.
  Interventions: Behavioral: Usual diet

INTERVENTIONS:
Behavioral: Low-energy dense diet — Subjects will follow time-restricted eating of a low energy dense diet
  Arms: Low energy dense diet
Behavioral: Usual diet — Subjects will follow time-restricted eating of the usual diet
  Arms: Usual diet

SUMMARY:
The goal of this randomized controlled trial is to test the effect of time-restricted eating (14-hour fast, 10-hour eating window) of a low-energy dense diet (reduced calories per gram of food) in older adults with obesity and insulin resistance. The study aims to determine if modulating the energy density of the diet reduces:

1. Insulin resistance and
2. Body weight.

Researchers will compare the groups:

1. Following time-restricted eating and given a diet reduced in energy density or
2. Following time-restricted eating and given a diet typically consumed in this population

DETAILED DESCRIPTION:
The study is an eight-week randomized controlled double-blinded clinical trial. Participants will follow time-restricted eating (14-hour fast, 10-hour eating window), and will be randomized to a diet low in energy density or the usual diet. Meals will be prepared in a metabolic kitchen and dispensed to participants. Dietitians will monitor dietary compliance. A blood sample will be drawn and body weight will be measured before starting the intervention and after completing it.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) ≥ 30kg/m2.
2. Mini-Mental State Examination (MMSE) > 25
3. Geriatric Depression Scale-15 (GDS-15) < 9
4. Homeostatic model assessment of insulin resistance (HOMA-IR) ≥ 3.

Exclusion Criteria:

1. Diagnosis of Type 2 diabetes received more than five years ago
2. Diagnosis of type 1 diabetes
3. Evidence of clinically significant renal dysfunction or disease
4. History of malignancy during the past five years
5. Being treated with systemic steroids, olanzapine, or clozapine
6. Being treated with prescription medications for obesity
7. Being treated with thiazolidinediones, glucagon-like-receptor agonists, Dipeptidyl Peptidase IV inhibitors, and insulin
8. Weight change > 3 kg in the preceding three months
9. Any disease or condition that precludes testing of the study outcomes or makes it unsafe to consume the foods being tested in the study, or subjects are otherwise deemed to be unsuitable for participation in the study (determined by the investigative team)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-29 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
Brain Insulin Resistance | 8 weeks
  Phosphorylation of serine 312 on insulin receptor substrate 1 in plasma neural-derived exosomes
Ketones | 8 weeks
  Ketones
Body weight | 8 weeks
  Body weight
Peripheral insulin resistance | 8 weeks
  Homeostasis model assessment of insulin resistance (HOMA-IR)

CONTACTS AND LOCATIONS:
Overall Officials: Candida Rebello, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No